CLINICAL TRIAL: NCT02066324
Title: Urine Sample Collection From Patients With Fibrodysplasia Ossificans Progressiva (FOP) for Biomarker Analysis
Brief Title: Urine Sample Collection From FOP Patients
Acronym: FOP
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CPJMR0062203
Record Dates: First submitted 2014-02-05; First posted 2014-02-19 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Fibrodysplasia Ossificans Progressiva
MeSH Terms: conditions — Myositis Ossificans

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect urine samples from patients with fibrodysplasia ossificans progressiva (FOP) for the assessment of biomarkers related to disease, disease progression and for prediction of flare-ups of the disease. Disease related biomarkers in these patients are currently unknown. This study aims to support the development of novel therapy/ies for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 5 and ≤ 35 years of age with a diagnosis of FOP.
* Physically able to provide first-morning urine sample of at least 30 mL
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* About half of the patients enrolled should have a flare-up, which is defined as an acute exacerbation of disease activity characterized by two or more of the following symptoms: pain, swelling, decreased range of motion, impaired function

Exclusion Criteria:

* Diagnosis of diabetes
* Diagnosis of other systemic inflammatory disorder (juvenile idiopathic arthritis, systemic lupus erythematosus, etc.)
* Diagnosis of cancer other than nonmelanomatous skin cancer.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Fibrodysplasia Ossificans Progressiva.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Analysis of pre-defined biomarker FGF2 | 3 months
  The objective of this study is to collect urine samples from patients with FOP over a time period covering ideally quiescent disease status and progression through a flare-up for biomarker analysis
Analysis of pre-defined biomarker WEGF | 3 months
  The objective of this study is to collect urine samples from patients with FOP over a time period covering ideally quiescent disease status and progression through a flare-up for biomarker analysis
Analysis of microRNAs | 3 months
  The objective of this study is to collect urine samples from patients with FOP over a time period covering ideally quiescent disease status and progression through a flare-up for biomarker analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Philadelphia, Pennsylvania, United States